CLINICAL TRIAL: NCT04867395
Title: A Multi-Phase Study Examining Hospital to Home Transitions for Children With Medical Complexity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-00180
Record Dates: First submitted 2021-04-28; First posted 2021-04-30 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Children With Medical Complexity (CMC)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): 75 participants will receive standard care, consisting of verbal discharge counseling given by doctors and nurses supplemented by written instructions (all unstandardized).
- Intervention group (Experimental): 75 participants will be randomized to receive behavioral intervention, consisting of discharge counseling using the health literacy-informed discharge instructions
  Interventions: Behavioral: HELPix Care Plan

INTERVENTIONS:
Behavioral: HELPix Care Plan — A web application tool for CMC - Health literacy-informed, disease and medication-specific, standardized discharge instructions that will: 1) facilitate plain language provider/parent communication at hospital discharge and 2) act as "stand-alone" handouts that parents can use at home.
  Arms: Intervention group

SUMMARY:
The overarching objective of this study is to make it easier for parents of children with medical complexity (CMC) to take care of their children after discharge home from the hospital and reduce the chance of post-hospitalization morbidity (meaning bad outcomes such as readmissions) after discharge. CMC, or those with multiple chronic conditions, progressive conditions, or technology dependence, are at high risk for post-hospitalization morbidity.

DETAILED DESCRIPTION:
This study will take place in 3 phases at 2 sites: Bellevue Hospital Center (BHC) and Hassenfeld Children's Hospital (HCH). Parents of CMC with a prior or current admission will be recruited at these two sites, as well as pediatricians who care for these children in the inpatient setting for the following 3 aims:

* In Aim 1, parents of CMC and pediatricians will be interviewed to understand their views on what makes it challenging, and what can make it easier, for parents to understand and follow the instructions they get from the hospital about how to take care of their CMC after leaving the hospital. The study team will also ask pediatricians what may make it difficult to provide relevant education to families.
* In Aim 2, a tool will be designed to make it easier for parents to understand and follow the discharge instructions for their CMC. The study team will use structure of existing tool, findings from Aim 1, and extensive interviews and testing of the tool with parents and pediatricians as the new tool is designed.
* In Aim 3, a randomized controlled trial (RCT) will be conducted to study the impact of the tool on parent comprehension and adherence (or how well they can follow) their child's discharge instructions, as well as its impact on post-discharge morbidity (such as readmissions and emergency department visits). Parents will be randomized to either receive usual hospital care and instructions or the intervention/tool (in addition to the usual care and instructions). The study team will also ask parents who receive the intervention about its usability.

ELIGIBILITY:
Inclusion Criteria:

Parents

* English or Spanish-speaking
* Parent or legal guardian and primary caregiver of child who has medical complexity (defined by significant chronic conditions in ≥2 body systems, progressive conditions associated with decreased life expectancy, dependence on technology for >6 months [e.g., respiratory equipment, central lines, feeding tubes], or progressive/metastatic malignancies) who was admitted to the acute or intensive care units
* The individual's child is ≤18 years old
* The individual's child was discharged home or is expected be discharged home on ≥1 daily medication.
* Willingness to be randomized to intervention group
* Willingness and ability to participate in study procedures

Exclusion Criteria:

Parents

* Caregiver <18 years old
* Poor visual acuity (<20/50 corrected on Rosenbaum screener for in-person recruitment; by subject report for phone recruitment)
* Self-reported hearing difficulty
* Previously enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Parent Comprehension of Discharge Instructions | Visit 2 (Day 0-1)
  The proportion of parents making errors in comprehension of their child's discharge instructions will be assessed. The visit will consist of a structured survey. Parents will be asked open-ended questions about their child's discharge instructions for their medications, appointments , return precautions , restrictions , equipment. Parents will be encouraged to use their written instructions when answering survey questions. The total proportion of parents making comprehension errors in an individual domain and across domains will be calculated. Errors in domains are defined by parent report of not following instructions properly. Comprehension in a given domain will be dichotomized into no errors vs. ≥1 error
Parent Adherence to Discharge Instructions | Visits 3-4 (Days 1-45)
  The proportion of parents making errors in adherence to their child's discharge instructions will be assessed with a structured survey. Parents will be asked open ended questions about their child's discharge instructions for their medications, appointments attended, return precautions, restrictions being followed, and equipment. Parents will be encouraged to use their written instructions when answering questions. Parents will be asked to measure out any liquid medications using a standard medication bottle as they would measure them at home.The total proportion of parents making adherence errors in an individual domain and across domains will be calculated.Medication dosing errors will be defined by >20% deviation from the prescribed dose for ≥1 medication as assessed by visual inspection as part of in-person dosing assessment. Appointment attendance errors will be defined by missing ≥1 scheduled appointment after discharge.
Number of CMC with any type of post-discharge morbidity | Visit 4 (Day 30-45)
  The total proportion of children with medical complexity (CMC) with any type of post-discharge morbidity (30-day readmissions, ED visits, outpatient visits, adverse drug events, surgical complications, infections) within 30 days of discharge will be calculated. Subjects will be dichotomized into those with no post-discharge morbidity vs. ≥1 type of postdischarge morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander F Glick, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to alexander.glick@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.